CLINICAL TRIAL: NCT00632333
Title: Phase I Study of Chemoradiation Therapy With Epitope Peptide Vaccine Therapy in Treating Patients With Unresectable, Advanced or Recurrent Esophageal Cancer
Brief Title: Combination of Chemoradiation Therapy and Epitope Peptide Vaccine Therapy in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teikyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Surgery, Teikyo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR07-079
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2009-09

CONDITIONS: Esophageal Cancer
Keywords: Epitope peptide; Vaccination; Chemoradiation; Esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — LY6K protein, human; Receptor Protein-Tyrosine Kinases; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: URLC10, TTK, KOC1, VEGFR1, VEGFR2, cisplatin, fluorouracil

INTERVENTIONS:
Biological: URLC10, TTK, KOC1, VEGFR1, VEGFR2, cisplatin, fluorouracil — Escalating dose of multiple peptides (URLC10, TTK, KOC1 VEGFR1, and VEGFR2) emulsified with Montanide ISA51 will be administered by subcutaneous injection on days 15, 22, 28 and 35 of treatment cycle. Doses of each peptide are planning 0.5mg, 1mg and 3mg/body. Chemotherapy plus radiation therapy will be done as follows: fluorouracil (400mg/m2) on day1-5 and 8-12, cisplatin (40mg/m2) on days 1 and 8, radiation (2Gy) on days 1-5, 8-12 and 15-19. Two cycles of combination of chemoradiation therapy and epitope peptide vaccine therapy will be done.
  Other Names: CDDP; 5-FU

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of multiple peptides (URLC10, TTK, KOC1 VEGFR1, and VEGFR2) emulsified with Montanide ISA51 in combination with chemotherapy (CDDP, 5-FU) plus radiation therapy in treating patients with unresectable, advanced or recurrent esophageal cancer.

DETAILED DESCRIPTION:
Up-regulated ling cancer 10 (URLC10), TTK protein kinase (TTK) and K homology domain containing protein over expressed in cancer (KOC1) were identified as new targets of tumor associated antigens using cDNA microarray technologies combined with the expression profiles of normal and cancer tissues. Furthermore, anti-angiogenic therapy is now considered to be one of promising approaches for treating cancer. Vascular endothelial growth factor receptor 1 (VEGFR1) and vascular endothelial growth factor receptor 2 (VEGFR2) are essential targets for tumor angiogenesis. Epitope peptides for these targets are able to induce cytotoxic T lymphocytes (CTL) restricted to HLA-A *2402 in vivo. On the other hand, chemotherapy (CDDP, 5-FU) plus radiation therapy has been to be a standard treatment for unresectable advanced esophageal cancer. In this clinical trial, we evaluate the safety and immune responses of different doses of multiple peptides (URLC10, TTK, KOC1, VEGFR1, and VEGFR 2) emulsified with Montanide ISA 51 in combination with chemotherapy (CDDP, 5-FU) plus radiation therapy in treating patients with unresectable, advanced or recurrent esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have unresectable, locally advanced, recurrent or metastatic disease of esophageal cancer.
2. measurable disease by CT scan
3. ECOG performance status of 0 to 2
4. Expected survival of at lease 3months
5. Patients must be HLA-A2402
6. Laboratory values as follow:

   * WBC > 2000/mm3,
   * Platelet count > 75000/mm3,
   * Total bilirubin < 1.5 x the institutional normal upper limits,
   * Creatinine < 1.5 x the institutional normal upper limits,
   * AST. ALT. ALP < 2.5 x the institutional normal upper limits
7. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential:Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Active or uncontrolled infection
4. Prior chemotherapy,radiation therapy or immunotherapy within 4 weeks
5. Concurrent treatment with steroid or immunosuppressing agent
6. Patient with peptic ulcer disease
7. Active or uncontrolled other malignancy
8. Other malignancy within 5 years prior to entry into the study, expect for treated non-melanoma skin cancer and cervical carcinoma in situ
9. Disease to the central nervous system
10. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Safety(toxicities as assessed by NCI CTCAE version3) | 3 months

SECONDARY OUTCOMES:
Peptide specific CTL induction | 3 months
DTH to peptide | 3 months
Changes in levels of regulatory T cells | 3 months
Objective response rate as assessed by RECIST criteria | 1 year
Time to progression | 1 year
survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kota Okinaga, MD, PhD, Study Chair — Teikyo University , Department Surgery
Locations (1):
- Teikyo University, 2-11-1 Kaga Itabashi-ku, Tokyo, Japan

REFERENCES:
- [Background] Yildirim Z, Kotuk M, Iraz M, Kuku I, Ulu R, Armutcu F, Ozen S. Attenuation of bleomycin-induced lung fibrosis by oral sulfhydryl containing antioxidants in rats: erdosteine and N-acetylcysteine. Pulm Pharmacol Ther. 2005;18(5):367-73. doi: 10.1016/j.pupt.2005.02.001. Epub 2005 Mar 23. PMID 15939316
- [Background] Li Y, Wang MN, Li H, King KD, Bassi R, Sun H, Santiago A, Hooper AT, Bohlen P, Hicklin DJ. Active immunization against the vascular endothelial growth factor receptor flk1 inhibits tumor angiogenesis and metastasis. J Exp Med. 2002 Jun 17;195(12):1575-84. doi: 10.1084/jem.20020072. PMID 12070285
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Date Y, Kimura A, Kato H, Sasazuki T. DNA typing of the HLA-A gene: population study and identification of four new alleles in Japanese. Tissue Antigens. 1996 Feb;47(2):93-101. doi: 10.1111/j.1399-0039.1996.tb02520.x. PMID 8851721
- [Background] Correale P, Cusi MG, Del Vecchio MT, Aquino A, Prete SP, Tsang KY, Micheli L, Nencini C, La Placa M, Montagnani F, Terrosi C, Caraglia M, Formica V, Giorgi G, Bonmassar E, Francini G. Dendritic cell-mediated cross-presentation of antigens derived from colon carcinoma cells exposed to a highly cytotoxic multidrug regimen with gemcitabine, oxaliplatin, 5-fluorouracil, and leucovorin, elicits a powerful human antigen-specific CTL response with antitumor activity in vitro. J Immunol. 2005 Jul 15;175(2):820-8. doi: 10.4049/jimmunol.175.2.820. PMID 16002679
- [Background] Nakopoulou L, Stefanaki K, Panayotopoulou E, Giannopoulou I, Athanassiadou P, Gakiopoulou-Givalou H, Louvrou A. Expression of the vascular endothelial growth factor receptor-2/Flk-1 in breast carcinomas: correlation with proliferation. Hum Pathol. 2002 Sep;33(9):863-70. doi: 10.1053/hupa.2002.126879. PMID 12378509
- [Background] Suda T, Tsunoda T, Uchida N, Watanabe T, Hasegawa S, Satoh S, Ohgi S, Furukawa Y, Nakamura Y, Tahara H. Identification of secernin 1 as a novel immunotherapy target for gastric cancer using the expression profiles of cDNA microarray. Cancer Sci. 2006 May;97(5):411-9. doi: 10.1111/j.1349-7006.2006.00194.x. PMID 16630140
- [Background] Watanabe T, Suda T, Tsunoda T, Uchida N, Ura K, Kato T, Hasegawa S, Satoh S, Ohgi S, Tahara H, Furukawa Y, Nakamura Y. Identification of immunoglobulin superfamily 11 (IGSF11) as a novel target for cancer immunotherapy of gastrointestinal and hepatocellular carcinomas. Cancer Sci. 2005 Aug;96(8):498-506. doi: 10.1111/j.1349-7006.2005.00073.x. PMID 16108831
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Dudley ME, Schwarz SL, Spiess PJ, Wunderlich JR, Parkhurst MR, Kawakami Y, Seipp CA, Einhorn JH, White DE. Immunologic and therapeutic evaluation of a synthetic peptide vaccine for the treatment of patients with metastatic melanoma. Nat Med. 1998 Mar;4(3):321-7. doi: 10.1038/nm0398-321. PMID 9500606
- [Background] Ishida K, Ando N, Yamamoto S, Ide H, Shinoda M. Phase II study of cisplatin and 5-fluorouracil with concurrent radiotherapy in advanced squamous cell carcinoma of the esophagus: a Japan Esophageal Oncology Group (JEOG)/Japan Clinical Oncology Group trial (JCOG9516). Jpn J Clin Oncol. 2004 Oct;34(10):615-9. doi: 10.1093/jjco/hyh107. PMID 15591460
- [Background] Waters JS, Tait D, Cunningham D, Padhani AR, Hill ME, Falk S, Lofts F, Norman A, Oates J, Hill A. A multicentre phase II trial of primary chemotherapy with cisplatin and protracted venous infusion 5-fluorouracil followed by chemoradiation in patients with carcinoma of the oesophagus. Ann Oncol. 2002 Nov;13(11):1763-70. doi: 10.1093/annonc/mdf301. PMID 12419749
- [Background] Marchand M, van Baren N, Weynants P, Brichard V, Dreno B, Tessier MH, Rankin E, Parmiani G, Arienti F, Humblet Y, Bourlond A, Vanwijck R, Lienard D, Beauduin M, Dietrich PY, Russo V, Kerger J, Masucci G, Jager E, De Greve J, Atzpodien J, Brasseur F, Coulie PG, van der Bruggen P, Boon T. Tumor regressions observed in patients with metastatic melanoma treated with an antigenic peptide encoded by gene MAGE-3 and presented by HLA-A1. Int J Cancer. 1999 Jan 18;80(2):219-30. doi: 10.1002/(sici)1097-0215(19990118)80:23.0.co;2-s. PMID 9935203
- [Derived] Iinuma H, Fukushima R, Inaba T, Tamura J, Inoue T, Ogawa E, Horikawa M, Ikeda Y, Matsutani N, Takeda K, Yoshida K, Tsunoda T, Ikeda T, Nakamura Y, Okinaga K. Phase I clinical study of multiple epitope peptide vaccine combined with chemoradiation therapy in esophageal cancer patients. J Transl Med. 2014 Apr 3;12:84. doi: 10.1186/1479-5876-12-84. PMID 24708624